CLINICAL TRIAL: NCT04008186
Title: A Phase 1, Open-Label, 4-Part, Drug-Drug Interaction Study With Omaveloxolone in Healthy Subjects
Brief Title: A Clinical Drug-Drug Interaction (DDI) Study With Omaveloxolone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 408-C-1806
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adult Subjects
Keywords: RTA 408; RTA 408 capsules; omaveloxolone; omaveloxolone capsules; DDI
MeSH Terms: interventions — omaveloxolone; Midazolam; repaglinide; Metformin; Tablets; Rosuvastatin Calcium; Digoxin; Gemfibrozil; Itraconazole; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Omaveloxolone and Multiple Drugs (Part 1) (Experimental): Single oral doses of 2 mg midazolam, 1 mg repaglinide, 500 mg metformin, and a 10 mg rosuvastatin/0.25 mg digoxin cocktail on Days 1, 2, 3, and 5, respectively, and 18, 19, 20, and 22, respectively. Oral doses of 150 mg omaveloxolone on Days 12 to 27
  Interventions: Drug: Omaveloxolone; Drug: Midazolam oral solution; Drug: Repaglinide 1 MG; Drug: MetFORMIN 500 Mg Oral Tablet; Drug: Rosuvastatin; Drug: Digoxin tablet
- Omaveloxolone & Gemfibrozil (Part 2) (Experimental): Single oral doses of 150 mg omaveloxolone on Days 1 and 13. Oral doses of 600 mg gemfibrozil (twice daily) on Days 10 to 18
  Interventions: Drug: Omaveloxolone; Drug: Gemfibrozil Tablets
- Omaveloxolone and Itraconazole (Part 3) (Experimental): Single oral doses of 150 mg omaveloxolone on Days 1 and 13. Oral doses of 200 mg itraconazole on Days 10 to 18.
  Interventions: Drug: Omaveloxolone; Drug: Itraconazole capsule
- Omaveloxolone and Verapamil (Part 4) (Experimental): Single oral doses of 150 mg omaveloxolone on Days 1 and 13. Oral doses of 120 mg verapamil on Days 10 to 18.
  Interventions: Drug: Omaveloxolone; Drug: Verapamil Pill

INTERVENTIONS:
Drug: Omaveloxolone — 50 mg capsules
  Other Names: RTA 408
Drug: Midazolam oral solution — 2 mg/mL oral solution
  Arms: Omaveloxolone and Multiple Drugs (Part 1)
Drug: Repaglinide 1 MG — 1 mg tablet
  Arms: Omaveloxolone and Multiple Drugs (Part 1)
Drug: MetFORMIN 500 Mg Oral Tablet — 500 mg tablet
  Arms: Omaveloxolone and Multiple Drugs (Part 1)
Drug: Rosuvastatin — 10 mg tablet
  Arms: Omaveloxolone and Multiple Drugs (Part 1)
Drug: Digoxin tablet — 0.25 mg tablet
  Arms: Omaveloxolone and Multiple Drugs (Part 1)
Drug: Gemfibrozil Tablets — 600 mg tablet
  Arms: Omaveloxolone & Gemfibrozil (Part 2)
Drug: Itraconazole capsule — 100 mg capsule
  Arms: Omaveloxolone and Itraconazole (Part 3)
Drug: Verapamil Pill — 120 mg tablet
  Arms: Omaveloxolone and Verapamil (Part 4)

SUMMARY:
This study will assess the potential for clinical drug-drug interactions between omaveloxolone and a number of substrates and inhibitors of metabolic enzymes and drug transporters.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria at the Screening Visit unless otherwise stated:

* Males or females, of any race, between 18 and 55 years of age, inclusive.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, and a total body weight >50 kg.
* In good health.
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

Subjects will be excluded from the study if they satisfy any of the following criteria at the Screening visit, unless otherwise stated:

* Significant history or clinical manifestation of any major system disorder, as determined by the investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (cholecystectomy will not be allowed; uncomplicated appendectomy and hernia repair will be allowed).
* History of alcoholism or drug/chemical abuse within 2 years prior to Check in (Day 1).
* Abnormal laboratory values considered clinically significant by the investigator
* Clinically significant abnormal 12 lead ECGs
* Personal history of unexplained syncopal events, or family history of long QT syndrome or sudden unexplained death in a young person.
* Pulse rate <50 bpm or systolic blood pressure <110 mmHg.
* Alcohol consumption of >21 units per week for males and >14 units for females.
* Positive urine drug screen or positive alcohol breath test result or positive urine drug screen.
* Positive hepatitis panel and/or positive human immunodeficiency virus test. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days prior to dosing or 5 half lives (if known), whichever is longer, prior to dosing.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, unless deemed acceptable by the investigator (or designee).
* Have previously completed or withdrawn from this study or any other study investigating omaveloxolone, and have previously received the investigational product.
* Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Part 1 - Maximum concentration (Cmax) of probe drugs co-administered with omaveloxolone (midazolam, repaglinide, metformin, rosuvastatin, and digoxin) | 28 days
  Pharmacokinetics will be assessed by blood sampling for midazolam, repaglinide, metformin, rosuvastatin, and digoxin to determine maximum observed concentration (Cmax).
Part 1 - Area under the plasma concentration-time curve of (AUC) for probe drugs co-administered with omaveloxolone (midazolam, repaglinide, metformin, rosuvastatin, and digoxin) | 28 days
  Pharmacokinetics will be assessed by blood sampling for midazolam, repaglinide, metformin, rosuvastatin, and digoxin to determine area under the curve (AUC).
Part 2 - Maximum concentration (Cmax) of omaveloxolone | 23 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine maximum observed concentration (Cmax).
Part 2 - Area under the omaveloxolone concentration-time curve (AUC) | 23 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine area under the curve (AUC).
Part 3 - Maximum concentration (Cmax) of omaveloxolone | 23 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine maximum observed concentration (Cmax).
Part 3 - Area under the omaveloxolone concentration-time curve (AUC) | 28 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine area under the curve (AUC).
Part 4 - Maximum concentration (Cmax) of omaveloxolone | 23 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine maximum observed concentration (Cmax).
Part 4 - Area under the omaveloxolone concentration-time curve (AUC) | 28 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine area under the curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Zon, MD, Principal Investigator — Covance CRU Inc.
Locations (1):
- Covance Clinical Research Unit (CRU) Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/